CLINICAL TRIAL: NCT07244289
Title: Managed Access Programs for VAY736, Ianalumab
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CVAY736I12003M
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Primary Immune Thrombocytopenia; Sjögren's Syndrome
Keywords: MAP; Managed Access Program; VAY736; ianalumab; Primary Immune Thrombocytopenia (ITP); Sjögren's Syndrome (SjD); Expanded Access; Early Access; Compassionate use
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Sjogren's Syndrome | interventions — ianalumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ianalumab — Patients receive ianalumab
  Other Names: VAY736

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to VAY736, ianalumab

DETAILED DESCRIPTION:
* CVAY736I12003M - Available - Managed Access Program (MAP) Cohort Treatment Plan CVAY736I12003M to provide access to ianalumab (VAY736) for patients with Primary Immune Thrombocytopenia (ITP)
* CVAY736A1002M - Not yet available - Managed Access Program (MAP) Cohort Treatment Plan CVAY736A1002M to provide access to ianalumab for adult patients with Sjögren's disease

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enrol in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult